CLINICAL TRIAL: NCT00118560
Title: Perfusion and Metabolism During Exercise in Peripheral Arterial Disease
Brief Title: Exercise Training for Patients With Poor Leg Circulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Figoni, Stephen - Principal Investigator, Department of Veterans Affairs
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: B3644P
Record Dates: First submitted 2005-06-30; First posted 2005-07-11 (Estimated); Last update posted 2011-03-17 (Estimated); Status verified 2011-03

CONDITIONS: Diabetes Mellitus, Type 2; Intermittent Claudication
Keywords: Collateral Circulation; Exercise Therapy; Microcirculation; Oxygen; Positron-emission tomography; Walking
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Intermittent Claudication | interventions — Exercise

ARMS (1):
- 1 (Experimental): treadmill walking and calf exercise
  Interventions: Behavioral: Physical exercise; Behavioral: Physical walking

INTERVENTIONS:
Behavioral: Physical exercise — treadmill walking
Behavioral: Physical walking — calf muscle exercise

SUMMARY:
The purposes of this pilot project are to (a) determine changes in calf muscle blood flow and energy supply resulting from calf muscle exercise, and (b) to determine changes in these variables resulting from exercise training (walking and calf muscle exercise). This is a pilot study to prepare for a larger project in the future. Exercise and exercise training should increase blood flow and energy supply to the calf muscles.

DETAILED DESCRIPTION:
Specific Objectives: 1.Develop an appropriate graded calf exercise test protocol for evaluating perfusion and metabolism during exercise in subjects with peripheral arterial disease (PAD), 2.compare perfusion in gastroc-soleus and tibialis anterior muscles during exercise and recovery from exercise, and to compare metabolism in those muscles during exercise, 3.compare the perfusion during exercise and recovery between groups with and without PAD, and to compare metabolism during exercise between groups with and without PAD, 4.estimate sample sizes and effect sizes for a future clinical trial to determine the efficacy of walking and calf muscle exercise training for improving calf muscle perfusion and metabolism. 5.determine the sensitivity and specificity of the PET exercise test in classifying subjects into groups with or without PAD, and 6. determine the test-retest reliability coefficients of perfusion and metabolic measures.

Two groups of subjects will participate in this study. Group I (n=25 subjects with PAD) will undergo two sets of assessments. Each assessment will consist of completing three questionnaires, two exercise tests, and one PET scan session. Additionally, they will receive one MRI of the legs. Then they will participate in a three-month exercise training intervention consisting of treadmill walking and calf muscle exercise. Finally, they will repeat one set of assessments (listed above with MRI). Group II (n=25 healthy control subjects) will undergo two sets of assessments. Each assessment will consist of three questionnaires, two submaximal exercise tests, one MRI, and one PET scan session (no exercise tests). Additionally they will receive only one MRI. They will not participate in an exercise training intervention.

Experimental Design The project is a pilot study that is both cross-sectional and longitudinal in nature. The initial baseline measurement sessions will allow comparisons of acute perfusion and metabolic physiologic responses between two groups of subjects (with and without PAD). Duplicate testing for each subject will allow assessment of the test-retest reliability of the measurements. The PAD subjects' perfusion and metabolic responses will be assessed again after three months of exercise training (walking and calf muscle exercise). While not a definitive clinical trial of the exercise training intervention, the results should provide estimates of sample and effect sizes to design a more definitive future clinical trial.

Subjects Recruitment and Sampling: Fifty different subjects (N=50) will participate in the project, reflecting the available veteran patient population. The sample will include primarily men, of any age and ethnicity. Twenty-five subjects will have PAD and will be identified and recruited via convenience sampling primarily from the Physical Medicine and Rehabilitation (PM&R) Outpatient Clinic, Diabetes Clinic, and Peripheral Vascular Clinic at the VA West Los Angeles Healthcare Center (VAWLAHC). Other participants may be recruited from other VA Greater Los Angeles Healthcare System locations, specifically the Los Angeles Ambulatory Care Center and the Sepulveda Ambulatory Care Center. Twenty-five "normal" healthy control subjects will be recruited via convenience sampling from well veterans and the general community; the two groups will be matched on gender and age. We plan to enroll 25 subjects with PAD for the three-month exercise training intervention.

Screening and Consent: Research staff will recruit and interview prospective subjects. Prospective subjects who meet all initial inclusion and exclusion criteria will be requested to review and sign the IRB-approved informed consent form and will be enrolled in the project. A physician will physically examine prospective subjects and provide medical clearance prior to participation.

Assessments and Measurements

After screening and consent, the assessment process will progress in four phases:

1. Questionnaires to evaluate walking impairment, physical activity, and general health. The information will be used to better characterize the study groups.
2. Exercise tolerance testing to demonstrate claudication symptoms in PAD subjects during both treadmill walking and calf muscle exercise and to assess functional changes resulting from training. The control subjects will also perform the exercise tests, but these tests will be submaximal and without pain. The data will be used for comparison to the data from PAD subjects.
3. Magnetic Resonance Imaging (MRI) of the legs to measure popliteal artery diameter and document locations of individual muscles and muscle groups.
4. PET-exercise testing to measure muscle perfusion and glucose metabolism during calf muscle exercise and recovery.

ELIGIBILITY:
Inclusion Criteria:

Group I (n=25 PAD patients). This sample will represent the population of veterans with PAD with mild mobility impairment secondary to intermittent claudication in the gastrocsoleus muscles.

Inclusion Criteria for PAD Subjects:

* diagnosis of PAD (acute or chronic occlusive arterial disease), with or without diabetes mellitus
* positive Edinburgh Claudication Questionnaire
* Fontaine stage IIa only (mild claudication, walking distance > 200 feet (one-half block)
* ambulatory, without assistive devices
* calf muscle claudication within 10 minutes of treadmill walking and calf muscle exercise

Group II (n=25 normal control/reference subjects). This reference sample will represent the population of adults without PAD and related problems. They will undergo the PET-exercise testing for perfusion and glucose metabolism measurements, but will not perform the exercise training intervention.

Inclusion Criteria for Controls:

* healthy adults, matched by age and sex to PAD subjects

Exclusion Criteria:

Exclusion Criteria for PAD and Control Subjects

* PAD secondary to Buerger's disease, autoimmune arteritis, fibromuscular dysplasia, chronic and repetitive occupational trauma, venous stasis, hypercoagulability disorder, or arterial embolic disease.
* inability to perform ankle dorsi and plantar flexion exercise
* cigarette smoking within last 6 months
* severe claudication, leg rest pain, skin ulceration, necrosis or gangrene (Fontaine stage >= IIa)
* poorly controlled diabetes mellitus (bA1c >= 9%)
* poorly controlled hypertension (resting BP > 140/90 mmHg)
* Raynaud's syndrome
* changes in prescribed cardiovascular medications within the past 6 months
* exertional angina, dyspnea, fatigue, or dizziness
* severe coronary artery disease
* congestive heart failure
* severe COPD
* exercise intolerance limited by leg pain of nonvascular origin (e.g., arthritis, orthopedic pain)
* transmetatarsal or more proximal lower-extremity amputation
* nonambulatory in the last 6 months
* severe leg weakness preventing leg exercise
* surgery related to PAD during preceding 3 months
* myocardial infarction within preceding 3 months
* unstable claudication symptoms during preceding 3 months
* terminal disease with < 6 months prognosis
* dementia (Minimental score < 24) (Folstein et al., 1975)
* pregnancy (Females of childbearing potential will be given a pregnancy test prior to acceptance into the study.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2005-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
maximal exercise times on treadmill and calf ergometer | baseline and after 3 months of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Stephen F. Figoni, Principal Investigator — VA Greater Los Angeles Healthcare System, West LA
Locations (1):
- VA Greater Los Angeles Healthcare System, West LA, West Los Angeles, California, United States

REFERENCES:
- [Result] Figoni SF, Kunkel CF, Scremin AM, Scremin OU, Cohen B. Ergometric performance during exercise training in men with intermittent claudication. PM R. 2010 Jun;2(6):528-36. doi: 10.1016/j.pmrj.2010.03.009. PMID 20630439